CLINICAL TRIAL: NCT03574181
Title: Calibration Study of a Wearable Noninvasive Blood Alcohol Monitor
Brief Title: Calibration Study of a Blood Alcohol Level Smart Watch
Status: Terminated | Type: Observational
Why Stopped: Extensive changes to the watch design would be needed to produce a robust device.
Sponsor: Boston Medical Center (Other)
Collaborators: KWJ Engineering (Industry); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Eric Devine, Assistant Professor, Dept of Psychiatry, Boston Medical Center
Other Study IDs: H-36914; R44AA024651-02 (NIH)
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Alcohol Drinking
Keywords: Wrist watch blood alcohol level; Blood alcohol; Objective alcohol measure
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Floors and Floorcoverings

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Smartwatch to measure Blood Alcohol Level (BAL) — Subjects will wear a wristwatch with a sensor that measures blood alcohol level during a 1-hour period of consuming alcohol followed by a 5 hour observation period.

SUMMARY:
This trial is designed to test the accuracy of a wristwatch blood alcohol level monitor relative to alcohol breath testing. An established human laboratory self-administration procedure will be followed. Each subject will complete 2 clinic visits over a period of up to 21 days of participation. Study participation is comprised of a baseline assessment to determine eligibility and an alcohol self-administration trial to test the accuracy of the wrist watch blood alcohol level. Subjects will be recruited in two phases of 9 subjects each. The first phase will be conducted to validate a prototype of the wrist watch. The second phase will be conducted to validate a pre-production consumer model of the blood alcohol wrist watch.

DETAILED DESCRIPTION:
In this proposed study, the objective is to further demonstrate the reliability of this printed electrochemical gas sensor in the form of a wearable device. This demonstration of reliability among human subjects is an essential part of product development. The monitor will be in a wristband or watch form, similar to a smart watch. This device will be modern, attractive and comfortable. It will also have smart watch features including measuring key physiological parameters (e.g., pulse) and eventually will have connectivity to apps on smart phones and other devices. The aim of the work is to provide a new, noninvasive transdermal alcohol monitor into the market. The transdermal alcohol monitoring market has few wearable products available and innovation has been lacking in this field. This new product will take advantage of current trends in wearable technology. As the public becomes more comfortable with wearable sensors, the blood alcohol monitor will become popular with people interested in health and fitness who want to track their alcohol intake. The product will provide a new, highly reliable and sensitive method for tracking blood alcohol level. This may be particularly beneficial to individuals who seek to reduce the risk of alcohol use by limiting peak blood alcohol level. If successful, this technology could be adopted in many areas including clinical and medical treatment, employee wellness programs, alcohol clinical trials, and as part of brief interventions that target at-risk drinkers.

The specific objective of this study is to determine whether the printed electrochemical gas sensor designed to measure blood alcohol level will be sensitive and reliable when compared to a standard measure of blood alcohol level taken by a breathalyzer. If this sensor proves sensitive to changes in blood alcohol level and can reliably measure blood alcohol level relative to a "gold standard" method, there are significant opportunities to use this technology in consumer health applications and clinical research.

ELIGIBILITY:
Inclusion Criteria:

1. 21-55 years of age.
2. Can provide proof of age with state or federal picture Identification.
3. Consumes an average of ≥7 standard drinks per week (women) or ≥14 drinks per week (men) over the 28 days prior to consent.
4. Has consumed at least 4 standard drinks on a single day on at least two days in the past 28 days prior to consent.
5. Has a blood alcohol level = 0.000 at time of consent.
6. Is able to understand and provide written informed consent.
7. Body weight ≥ 120 lbs and ≤ 250 pounds
8. Subjects can speak and understand English

Exclusion Criteria:

1. Currently seeking treatment for alcohol problems or purposefully abstaining from alcohol in an attempt to cut back or quit drinking.
2. Clinical Institute Withdrawal Assessment at ≥10.
3. Meets DSM-5 diagnosis of current major depression, bipolar disorder, schizophrenia, bulimia/anorexia, dementia, or a substance use disorder other than alcohol, nicotine, marijuana, or caffeine
4. If female, pregnant or nursing.
5. If female, does not agree to use an accepted form of birth control
6. Has medical or mental condition for which further alcohol exposure at the planned dose range would be contraindicated.
7. Taking medication for which drinking would be contraindicated.
8. Clinically significant abnormal ECG.
9. AST or ALT ≥ 3x the upper limit of normal.
10. Current risk of suicidality.
11. Has taken medications that are used to treat AUD in the past 90 days.
12. Has received alcohol counseling or other non-pharmacologic intervention to treat alcohol use disorder in the past 90 days.
13. Has urine toxicology results positive for cocaine, opioids, amphetamines, buprenorphine, methadone, or methamphetamines.
14. Smokes greater than 5 cigarettes per day.
15. Unable to comfortably abstain from nicotine for a period of 8 hours.
16. Wearing cologne, perfume, aftershave or any other scented oil or alcohol-based beauty product on the day of the Alcohol Lab Visit.
17. Has dietary restrictions that would preclude participating.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Moderate (non-problem) drinking healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Devine, PhD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Psychiatry Research Center, Clinical Studies Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Transdermal Alcohol Sensor: Single-arm study. All eligible subjects consume two mixed drinks calibrated to raise their blood alcohol level to 0.05 g/dL over 60 minutes. Subjects are fitted with a transdermal alcohol sensor on each wrist. Breathalyzer measurements are taken every 15 minutes for a period of five hours following consumption of alcohol.
Period: Overall Study
Arm/Group | Transdermal Alcohol Sensor
Started | 9
Completed | 0
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Transdermal Alcohol Sensor: All eligible subjects consume two mixed drinks calibrated to raise their blood alcohol level to 0.05 g/dL over 60 minutes. Subjects are fitted with a transdermal alcohol sensor on each wrist. Breathalyzer measurements are taken every 15 minutes for a period of five hours following consumption of alcohol.
Arm/Group | Transdermal Alcohol Sensor
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 38 [22 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Breathalyzer and Wristwatch Sensor BAL Measurements
Description: Wristwatch sensor BAL is continuously measured for entirety of 6-hour alcohol self administration trial. BAL from breathalyzer (BrAC) is measured at 15-minute intervals throughout 6-hour alcohol self administration trial. The correlation between wristwatch transdermal BAL (TAC) and breathalyzer BAL (BrAC) for all subjects will be calculated.
Time Frame: 6 hours during alcohol self administration trial
Population: 6 of 9 participants were included in data analyses. Three participants were excluded from analyses due to inability to obtain TAC data from wristwatches during alcohol self administration trials.
Measure: Number; unit: coefficient of determination (R^2)
Groups:
- Transdermal Alcohol Sensor: Single-arm study. All eligible subjects consume two mixed drinks calibrated to raise their blood alcohol level to 0.05 g/dL over 60 minutes. Subjects are fitted with a transdermal alcohol sensor on each wrist. Breathalyzer measurements are taken every 15 minutes for a period of three hours following consumption of alcohol.
Arm/Group | Transdermal Alcohol Sensor
Number analyzed (Participants) | 6
coefficient of determination (R^2) | 0.3183

ADVERSE EVENTS:
Time Frame: up to 14 days
Description: The primary risks of this study were loss of confidentiality, discomfort with study procedures, overconsumption of alcohol, and interference with efforts for recovery from alcohol use disorder. These risks were adequately minimized by study design and adherence to the study protocol.
Arm/Group | Transdermal Alcohol Sensor
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
The large variability in response characteristics between individuals and the complexity of model development in the face of the large BrAC - TAC lag times presented challenges to further development and completion of phase 2 of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03574181/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT03574181/ICF_001.pdf